CLINICAL TRIAL: NCT06203002
Title: A Phase 2b, Dose-ranging, Randomized, Double-blind, PlacebO-controlled, Parallel-GRoup, MulticEnter Study in PatientS With Diabetic Peripheral Neuropathic Pain (PROGRESS)
Brief Title: A Dose-ranging Study in Patients With Diabetic Peripheral Neuropathic Pain (DPNP)
Acronym: PROGRESS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LX9211.1-204-DPN; LX9211.204-DPN (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2023-11-30; First posted 2024-01-12 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Diabetic Peripheral Neuropathic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LX9211 Low Dose (Experimental): LX9211 low dose, orally, once daily during a blinded treatment period.
  Interventions: Drug: LX9211 (blinded)
- LX9211 High Dose (Experimental): LX9211 high dose, orally, once daily during a blinded treatment period.
  Interventions: Drug: LX9211 (blinded)
- LX9211 High Dose Followed by Low Dose (Experimental): LX9211 high dose followed by LX9211 low dose, orally, once daily during a blinded treatment period.
  Interventions: Drug: LX9211 (blinded)
- LX9211 Placebo (Placebo Comparator): LX9211 matching placebo, orally, once daily during a blinded treatment period.
  Interventions: Drug: Placebo (blinded)

INTERVENTIONS:
Drug: Placebo (blinded) — LX9211 matching placebo tablets
  Arms: LX9211 Placebo
Drug: LX9211 (blinded) — LX9211 (blinded) tablets
  Arms: LX9211 High Dose; LX9211 High Dose Followed by Low Dose; LX9211 Low Dose

SUMMARY:
Evaluation of the efficacy of LX9211 compared to placebo in reducing DPNP. Please see study website: https://diabeticpainstudy.com/

ELIGIBILITY:
Inclusion Criteria:

1. Participant has given written informed consent to participate in the study in accordance with local regulations
2. Adult male and female participants ≥18 years of age at the Screening Visit
3. Body mass index ≥18.0 to ≤40.0 kilogram per meter square (kg/m^2) at Screening
4. Diagnosis of type 1 diabetes mellitus (T1DM) or type 2 diabetes mellitus (T2DM) with chronic DPNP, at Screening
5. Pain from DPNP present for at least 6 months prior to Screening
6. At the Screening Visit, glycosylated hemoglobin (A1C) must be ≤11%.
7. Stable regimen for the treatment of T1DM or T2DM for ≥3 months prior to Screening
8. Willing to adhere to the prohibitions and restrictions specified in the protocol.

Exclusion Criteria:

1. Presence of other painful conditions that may confound assessment or self-evaluation of DPNP
2. History of neurolytic or neurosurgical therapy for DPNP
3. Use of opioid medications for management of DPNP within the 2 months prior to the Screening Visit.
4. Use of prescription topical analgesics (eg, capsaicin) indicated for neuropathic pain within 3 months prior to Screening
5. Use of nonsteroidal anti-inflammatory drugs (NSAIDs) less than 2 weeks prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 8 in Average Daily Pain Score (ADPS) | Baseline, Week 8
  ADPS is based on the 11-point numerical rating scale (NRS) [0 (no pain) to 10 (worst imaginable pain)].

SECONDARY OUTCOMES:
Change from Baseline to Week 8 in Burning Pain | Baseline, Week 8
  Burning pain is based on the 11-point NRS (0 [no burning] to 10 [worst burning imaginable]).
Change from Baseline to Week 8 in Pain Interference on Sleep | Baseline, Week 8
  Pain interference on sleep is based on the 11-point NRS (0 [does not interfere] to 10 [completely interferes]).
Patient Global Impression of Change (PGIC) Score at Week 8 | Week 8
  The PGIC is a 7-point rating scale that assesses a participant's belief about the overall improvement experienced by the participant where 1=very much improved and 7=very much worse.
Change from Baseline to Week 8 in Total Neuropathic Pain Symptom Inventory (NPSI) Score | Baseline, Week 8
  NPSI total score is based on 5 subscales evaluating different symptoms of neuropathic pain, each evaluated on a scale of 0 (no pain) to 10 (worst pain). The total score ranges from 0 to 100. A higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Locations (108):
- United States (108):
  - Lexicon Investigational Site (128), Anniston, Alabama
  - Lexicon Investigational Site (222), Birmingham, Alabama
  - Lexicon Investigational Site (189), Daphne, Alabama
  - Lexicon Investigational Site (215), Guntersville, Alabama
  - Lexicon Investigational Site (115), Chandler, Arizona
  - Lexicon Investigational Site (195), Phoenix, Arizona
  - Lexicon Investigational Site (206), Scottsdale, Arizona
  - Lexicon Investigational Site (102), Tucson, Arizona
  - Lexicon Investigational Site (107), Anaheim, California
  - Lexicon Investigational Site (173), Canoga Park, California
  - Lexicon Investigational Site (179), Escondido, California
  - Lexicon Investigational Site (161), Fresno, California
  - Lexicon Investigational Site (112), Greenbrae, California
  - Lexicon Investigational Site (204), Huntington Beach, California
  - Lexicon Investigational Site (191), Inglewood, California
  - Lexicon Investigational Site (163), Lomita, California
  - Lexicon Investigational Site (169), Long Beach, California
  - Lexicon Investigational Site (111), Sacramento, California
  - Lexicon Investigational Site (126), Sacramento, California
  - Lexicon Investigational Site (129), San Diego, California
  - Lexicon Investigational Site (154), San Diego, California
  - Lexicon Investigational Site (124), Tustin, California
  - Lexicon Investigational Site (211), Vista, California
  - Lexicon Investigational Site (171), Walnut Creek, California
  - Lexicon Investigational Site (181), Walnut Creek, California
  - Lexicon Investigational Site (119), Brandon, Florida
  - Lexicon Investigational Site (194), Brandon, Florida
  - Lexicon Investigational Site (177), Daytona Beach, Florida
  - Lexicon Investigational Site (198), Fleming Island, Florida
  - Lexicon Investigational Site (109), Fort Myers, Florida
  - Lexicon Investigational Site (180), Hollywood, Florida
  - Lexicon Investigational Site (188), Jacksonville, Florida
  - Lexicon Investigational Site (164), Miami, Florida
  - Lexicon Investigational Site (105), New Port Richey, Florida
  - Lexicon Investigational Site (146), Orlando, Florida
  - Lexicon Investigational Site (144), Orlando, Florida
  - Lexicon Investigational Site (123), Ormond Beach, Florida
  - Lexicon Investigational Site (182), Plantation, Florida
  - Lexicon Investigational Site (133), The Villages, Florida
  - Lexicon Investigational Site (138), The Villages, Florida
  - Lexicon Investigational Site (131), Winter Haven, Florida
  - Lexicon Investigational Site (103), Winter Park, Florida
  - Lexicon Investigational Site (150), Atlanta, Georgia
  - Lexicon Investigational Site (151), Marietta, Georgia
  - Lexicon Investigational Site (172), Chicago, Illinois
  - Lexicon Investigational Site (132), Flossmoor, Illinois
  - Lexicon Investigational Site (185), El Dorado, Kansas
  - Lexicon Investigational Site (178), Newton, Kansas
  - Lexicon Investigational Site (186), Wichita, Kansas
  - Lexicon Investigational Site (213), Owensboro, Kentucky
  - Lexicon Investigational Site (170), New Orleans, Louisiana
  - Lexicon Investigational Site (190), New Orleans, Louisiana
  - Lexicon Investigational Site (121), Boston, Massachusetts
  - Lexicon Investigational Site (140), New Bedford, Massachusetts
  - Lexicon Investigational Site (225), Waltham, Massachusetts
  - Lexicon Investigational Site (125), Ann Arbor, Michigan
  - Lexicon Investigational Site (108), Dearborn, Michigan
  - Lexicon Investigational Site (139), Olive Branch, Mississippi
  - Lexicon Investigational Site (104), Hazelwood, Missouri
  - Lexicon Investigational Site (174), Kansas City, Missouri
  - Lexicon Investigational Site (184), Springfield, Missouri
  - Lexicon Investigational Site (156), St Louis, Missouri
  - Lexicon Investigational Site (116), Papillion, Nebraska
  - Lexicon Investigational Site (216), Las Vegas, Nevada
  - Lexicon Investigational Site (162), Las Vegas, Nevada
  - Lexicon Investigational Site (142), New York, New York
  - Lexicon Investigational Site (227), Rochester, New York
  - Lexicon Investigational Site (167), Schenectady, New York
  - Lexicon Investigational Site (122), Westfield, New York
  - Lexicon Investigational Site (110), Williamsville, New York
  - Lexicon Investigational Site (200), Asheville, North Carolina
  - Lexicon Investigational Site (209), Greensboro, North Carolina
  - Lexicon Investigational Site (212), Monroe, North Carolina
  - Lexicon Investigational Site (106), Morehead City, North Carolina
  - Lexicon Investigational Site (145), Winston-Salem, North Carolina
  - Lexicon Investigational Site (220), Beavercreek, Ohio
  - Lexicon Investigational Site (168), Dayton, Ohio
  - Lexicon Investigational Site (148), Norman, Oklahoma
  - Lexicon Investigational Site (210), Oklahoma City, Oklahoma
  - Lexicon Investigational Site (187), Eugene, Oregon
  - Lexicon Investigational Site (183), Charleston, South Carolina
  - Lexicon Investigational Site (201), Columbia, South Carolina
  - Lexicon Investigational Site (113), Greenville, South Carolina
  - Lexicon Investigational Site (205), North Charleston, South Carolina
  - Lexicon Investigational Site (202), Rock Hill, South Carolina
  - Lexicon Investigational Site (157), Summerville, South Carolina
  - Lexicon Investigational Site (160), Memphis, Tennessee
  - Lexicon Investigational Site (192), Austin, Texas
  - Lexicon Investigational Site (199), Baytown, Texas
  - Lexicon Investigational Site (193), Dallas, Texas
  - Lexicon Investigational Site (158), Dallas, Texas
  - Lexicon Investigational Site (153), Euless, Texas
  - Lexicon Investigational Site (114), Flower Mound, Texas
  - Lexicon Investigational Site (196), Harlingen, Texas
  - Lexicon Investigational Site (120), Houston, Texas
  - Lexicon Investigational Site (197), Houston, Texas
  - Lexicon Investigational Site (152), Houston, Texas
  - Lexicon Investigational Site (214), Katy, Texas
  - Lexicon Investigational Site (155), Lewisville, Texas
  - Lexicon Investigational Site (223), Mesquite, Texas
  - Lexicon Investigational Site (203), San Antonio, Texas
  - Lexicon Investigational Site (159), San Antonio, Texas
  - Lexicon Investigational Site (221), San Antonio, Texas
  - Lexicon Investigational Site (101), Salt Lake City, Utah
  - Lexicon Investigational Site (219), Salt Lake City, Utah
  - Lexicon Investigational Site (224), St. George, Utah
  - Lexicon Investigational Site (130), Manassas, Virginia
  - Lexicon Investigational Site (165), Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No